CLINICAL TRIAL: NCT05132114
Title: Large Loop Excision of the Transformation Zone (LLETZ) with Versus Without Intraoperative Application of Lugol's Iodine in Women with Cervical Dysplasia: a Prospective Randomized Trial
Brief Title: Large Loop Excision of the Transformation Zone (LLETZ) with Vs Without IntraOperative Application of Lugol's Iodine
Acronym: LLETZ-IOLI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Clemens Tempfer, Director, Department of Obstetrics and Gynecologiy, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LLETZ-IOLI-1
Record Dates: First submitted 2021-11-11; First posted 2021-11-24 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Cervical Dysplasia
Keywords: cervical dyslasia; LLETZ; LEEP; Lugol's iodine; conization
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Intervention Model Description: Prospective randomized trial with 2 groups (use vs not use of Lugol's iodine during LLETZ)
Who Masked: Participant
Masking Description: Participants are not aware of their treatment allocation in order not to influence patient reported outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): LLETZ (without intraoperative Lugol's iodine)
- Iodine group (Experimental): LLETZ after the intraoperative application of Lugol's iodine
  Interventions: Diagnostic Test: Lugol's iodine test

INTERVENTIONS:
Diagnostic Test: Lugol's iodine test — Intraoperative application of Lugol's iodine (i.e. staining of the cervix with Lugol's iodine solution)
  Arms: Iodine group

SUMMARY:
Cervical cancer is one of the most common cancers in women and one of the leading causes of death in women worldwide. Pre-cancerous lesions (dysplasias) are detected by the gynecologist's preventive smear test and can thus contribute to a 100% chance of cure if they are clarified by a colposcopic examination as part of the dysplasia consultation and, if necessary, surgically removed. Conization (= surgical removal of a cone of tissue from the cervix) is the method of choice for removing the diseased tissue. LLETZ conization (Large Loop Excision of the Transformation Zone) is the worldwide standard surgical procedure for conization. There is risk of local persistence of the precancerous lesion if the cervical dysplasia is not completely removed. To minimize this, the iodine test can be used. Here, a 5% iodine solution (so-called Lugol's solution) is dabbed onto the cervix uteri, resulting in an intense and characteristic brown staining of the healthy cervical epithelium. Sites without staining are termed iodine negative and may contain dysplastic cells. The strength of iodine testing lies in its high specificity, i.e., the reliable ability to exclude false-positive results. The purpose of intraoperative iodine staining is to select the resection line with a high degree of certainty in healthy (i.e., iodine-positive) tissue in order to reduce the rate of cervical dysplasia that is not completely removed (so-called non-in-sano resection, or R1 resection). Systematic survey data from the dysplasia units certified in Germany on the question of the use of intraoperative iodine testing in Germany are lacking, as is the literature as a whole. For example, the current S3 guideline of the German Society of Gynecology and Obstetrics on the diagnosis and treatment of cervical dysplasia (as of March 2020) names intraoperative iodine testing only as a possible option for performing LLETZ.

In this prospective, randomized study, the investigators aim to answer the question whether LLETZ performed with the help of an iodine test with selection of the resection line in the iodine-positive area leads to a lower rate of R1 resections compared to the standard LLETZ without iodine test.

DETAILED DESCRIPTION:
1. Background 1.1. HPV and dysplasias of the cervix uteri Human papillomaviruses (HPV) are the most common sexually transmitted pathogens worldwide. The prevalence in both male and female populations is high. Epidemiological estimates suggest that 85-91% of sexually active adults acquire at least one genital HPV infection by the age of 50, with approximately 95% of HPV infections being spontaneously eliminated within 2 years in terms of HPV immunological clearance. HPV preferentially infects the epithelial cells of the anogenital area and, through incorporation of HPV DNA into the host genome of the basal cells of the squamous epithelium of the cervix and subsequent expression of viral components, causes dysplastic changes in the cervical epithelium that, if left untreated, can develop into invasive carcinoma of the cervix (cervical carcinoma). Cervical carcinoma is the fourth most common cancer as well as the fourth leading cause of cancer-related death in women worldwide, responsible for 6.6% (570,000) of all new cancer cases and 7.5% (311,000) of cancer-related deaths in women in 2018. The precursor of squamous cell carcinoma of the uterine cervix (approximately 80% of all cervical cancers) is cervical intraepithelial neoplasia (CIN), which has three grades of expression (CIN1, CIN 2, and CIN 3). Compared with invasive cervical carcinoma, the incidence of precancerous lesions of the cervix uteri is much higher. It is estimated that approximately 100,000 women in Germany develop high-grade dysplasia (CIN2/CIN3) annually.

   1.2. Surgical treatment If precancerous lesions with the potential to develop into an invasive cervical tumor are detected, conization (= surgical removal of a cone of tissue from the cervix) is the method of choice for removing the diseased tissue. Worldwide standard as surgical procedure for conization is LLETZ-conization (Large Loop Excision of the Transformation Zone). In addition to the risk of local persistence of the precancerous lesion if the cervical dysplasia is incompletely removed, LLETZ also increases the risk of preterm birth in a subsequent pregnancy. This risk increases with increasing volume of removed tissue. To reduce or avoid the aforementioned complications, conization should be performed under colposcopic vision and as little healthy cervical tissue as possible should be removed. One method of LLETZ that is as tissue-conserving as possible is the intraoperative use of the so-called 'iodine test'.

   1.3. The iodine test For the identification of healthy squamous epithelium of the cervix uteri, the so-called Schiller's iodine test can be used, which has been part of the clinical routine in the context of colposcopy of cervical dysplasias for decades. In the iodine test, a 5% iodine solution (so-called Lugol's solution) is dabbed onto the cervix uteri, resulting in an intense and characteristic brown staining of the healthy cervical epithelium. Sites without staining are termed iodine negative and may contain dysplastic cells. The strength of iodine testing lies in its high specificity, i.e., the reliable ability to exclude false-positive results. Not all iodine-negative areas contain CIN, but iodine-positive areas are almost certainly healthy. In some centers, because of these characteristics of the iodine sample, it is used during LLETZ to define the resection line of LLETZ. The aim of this approach is to select the resection line with a high degree of certainty in healthy (i.e., iodine-positive) tissue in order to reduce the rate of cervical dysplasia that is not completely removed (so-called 'non-in-sano resection' or 'R1 resection'). Systematic survey data from the dysplasia units certified in Germany on the question of the use of intraoperative iodine testing in Germany are lacking. The current S3 guideline of the German Society of Gynecology and Obstetrics on the diagnosis and therapy of cervical dysplasia (as of March 2020) also refers to intraoperative iodine testing as a possible option for performing LLETZ. However, exact figures from controlled studies on the usefulness of iodine test-guided LLETZ are lacking in the literature (PubMed search on 10/15/2021; search terms: cervical dysplasia, colposcopy, Lugol's test, iodine test, Lugol's staining; LLETZ; LEEP; conization). At our certified dysplasia center, it is the decision of the respective surgeon whether an additional intraoperative iodine test is performed or not.
2. Aim of the study The aim of this study is to answer the question under prospective randomized conditions whether LLETZ performed with the aid of iodine assay with selection of the resection line in the iodine-positive region leads to a lower rate of R1 resections compared with standard LLETZ without iodine assay.

ELIGIBILITY:
Inclusion Criteria:

* Written consent
* Colposcopy performed preoperatively
* Histologically (by previously performed colposcopy) confirmed dysplasia (CIN 1, CIN 2 or CIN 3)
* Age >18 years

Exclusion Criteria:

* Pregnant patients
* Patients with insufficient knowledge of the German language
* Treatments already performed on the cervix uteri, in particular conization
* Blood coagulation disorders
* Taking blood thinning substances
* Iodine allergy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2022-01-17 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Rate of R1 resections | Specimen from surgery (result expected 1-2 days after surgery)
  The primary outcome parameter is the rate of R1 resections, defined as the presence of a CIN I, CIN II, or CIN III at the ectocervical and/or endocervical resection margin, as indicated in the histopathologic report.

SECONDARY OUTCOMES:
Cone mass | During surgery, immediately after the excision
  The weight of the cone specimen (measured in grams in the unfixed state)
Procedure duration | At surgery
  Duration of the procedure (from start until complete hemostasis is achieved)
Rate of complications | During surgery up to 14 days post surgery
  The occurring intra- and postoperative complications in a period within 14 days after surgery
Surgeon's rating of handling | Immediately after surgery
  The assessment of the surgeon's handling of the surgical technique (LLETZ with/without intraoperative iodine assay) (11-item numerical rating scale [NRS]; 0 = very cumbersome, 10 = very easy)
Surgeon's satisfaction | Immediately after surgery
  The surgeon's satisfaction with the course of the operation in general (11-item NRS; 0 = no satisfied at all, 10 = very satisfied)
Time to complete hemostasis | During surgery
  The time from start of electro-coagulation until complete hemostasis (seconds)
Blood loss | At surgery
  The intraoperative blood loss (measured as the difference between preoperative and 3-5 hours postoperative Hb levels).

CONTACTS AND LOCATIONS:
Overall Officials: Clemens B Tempfer, MD, MBA, Principal Investigator — Ruhr-Universität Bochum / Marien Hospital Herne
Locations (1):
- Marien Hospital Herne, Herne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request made to the corresponding author. This includes individual participant data underlying the results presented here, after deidentification, as well as data dictionaries and the the study protocol. Data is available after publication, without a specific end date. Requesting investigators must show that their proposed use of the data has been approved by an independent review committee identified for this purpose.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After publication of the study results, no time limit.
Access Criteria: Reasonable request, approval of the intended study by an independent review committee identified for this purpose.

REFERENCES:
- [Background] Workowski KA, Bachmann LH, Chan PA, Johnston CM, Muzny CA, Park I, Reno H, Zenilman JM, Bolan GA. Sexually Transmitted Infections Treatment Guidelines, 2021. MMWR Recomm Rep. 2021 Jul 23;70(4):1-187. doi: 10.15585/mmwr.rr7004a1. PMID 34292926
- [Background] Chesson HW, Dunne EF, Hariri S, Markowitz LE. The estimated lifetime probability of acquiring human papillomavirus in the United States. Sex Transm Dis. 2014 Nov;41(11):660-4. doi: 10.1097/OLQ.0000000000000193. PMID 25299412
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Mathevet P, Chemali E, Roy M, Dargent D. Long-term outcome of a randomized study comparing three techniques of conization: cold knife, laser, and LEEP. Eur J Obstet Gynecol Reprod Biol. 2003 Feb 10;106(2):214-8. doi: 10.1016/s0301-2115(02)00245-2. PMID 12551795
- [Background] Bevis KS, Biggio JR. Cervical conization and the risk of preterm delivery. Am J Obstet Gynecol. 2011 Jul;205(1):19-27. doi: 10.1016/j.ajog.2011.01.003. Epub 2011 Feb 23. PMID 21345402
- [Background] Jin G, LanLan Z, Li C, Dan Z. Pregnancy outcome following loop electrosurgical excision procedure (LEEP) a systematic review and meta-analysis. Arch Gynecol Obstet. 2014 Jan;289(1):85-99. doi: 10.1007/s00404-013-2955-0. Epub 2013 Jul 11. PMID 23843155
- [Background] Khalid S, Dimitriou E, Conroy R, Paraskevaidis E, Kyrgiou M, Harrity C, Arbyn M, Prendiville W. The thickness and volume of LLETZ specimens can predict the relative risk of pregnancy-related morbidity. BJOG. 2012 May;119(6):685-91. doi: 10.1111/j.1471-0528.2011.03252.x. Epub 2012 Feb 14. PMID 22329499
- [Background] Shaco-Levy R, Eger G, Dreiher J, Benharroch D, Meirovitz M. Positive margin status in uterine cervix cone specimens is associated with persistent/recurrent high-grade dysplasia. Int J Gynecol Pathol. 2014 Jan;33(1):83-8. doi: 10.1097/PGP.0b013e3182763158. PMID 24300540
- [Background] Preaubert L, Gondry J, Mancini J, Chevreau J, Lamblin G, Atallah A, Lavoue V, Caradec C, Baldauf JJ, Bryand A, Henno S, Villeret J, Agostini A, Douvier S, Jarniat A, Riethmuller D, Mendel A, Brun JL, Rakotomahenina H, Carcopino X. Benefits of Direct Colposcopic Vision for Optimal LLETZ Procedure: A Prospective Multicenter Study. J Low Genit Tract Dis. 2016 Jan;20(1):15-21. doi: 10.1097/LGT.0000000000000156. PMID 26704328
- [Background] Kuhn W. [Colposcopy in the diagnosis of early cervical cancer]. Pathologe. 2011 Nov;32(6):497-504. doi: 10.1007/s00292-011-1480-9. German. PMID 21984389
- [Background] Hilal Z, Rezniczek GA, Alici F, Kumpernatz A, Dogan A, Alieva L, Tempfer CB. Loop electrosurgical excision procedure with or without intraoperative colposcopy: a randomized trial. Am J Obstet Gynecol. 2018 Oct;219(4):377.e1-377.e7. doi: 10.1016/j.ajog.2018.07.023. Epub 2018 Jul 29. PMID 30063903
- [Background] Rezniczek GA, Hecken JM, Rehman S, Dogan A, Tempfer CB, Hilal Z. Syringe or mask? Loop electrosurgical excision procedure under local or general anesthesia: a randomized trial. Am J Obstet Gynecol. 2020 Dec;223(6):888.e1-888.e9. doi: 10.1016/j.ajog.2020.06.041. Epub 2020 Jul 24. PMID 32585223
- [Background] Hilal Z, Rezniczek GA, El-Fizazi N, Tempfer CB. Large Loop Excision of the Transformation Zone Versus True Cone Biopsy Electrode Excision: A Randomized Trial. J Low Genit Tract Dis. 2017 Oct;21(4):272-278. doi: 10.1097/LGT.0000000000000329. PMID 28953118
- See also: German S3 Guidelines — https://www.leitlinienprogramm-onkologie.de/leitlinien/zervixkarzinom-praevention/